CLINICAL TRIAL: NCT01869062
Title: Clinical Assessment of the SonR Algorithm in the PARADYM RF SonR CRT-D by Echocardiography
Acronym: SonR-ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ICSY01
Record Dates: First submitted 2013-05-27; First posted 2013-06-05 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
Keywords: CRT
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: CRT-D device
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SonR CRT Optimization 'On' (Other): CRT-D device with the SonR optimization algorithm programmed being 'on'.
  Interventions: Device: SonR CRT Optimization 'On'
- SonR CRT Optimization 'Off' (Other): CRT-D device with the SonR optimization algorithm programmed being 'off' (Standard of Care).
  Interventions: Device: SonR CRT Optimization 'Off'

INTERVENTIONS:
Device: SonR CRT Optimization 'On' — Intervention: Implanted CRT-D device with the SonR optimization algorithm programmed being 'on'.
  Arms: SonR CRT Optimization 'On'
Device: SonR CRT Optimization 'Off' — Intervention: Implanted CRT-D device with the SonR optimization algorithm programmed being 'off' (Standard of Care).
  Arms: SonR CRT Optimization 'Off'

SUMMARY:
The main objective of the SONR-ECHO trial is to demonstrate that optimization of CRT parameters by SonR technology is able to increase the rate of CRT-D responders, based on significant LV reverse remodeling, as compared to Standard of Care settings.

This study will also evaluate the effectiveness of CRT-D SonR system as compared to Standard of care (SoC) programming methods in providing appropriate LV filling, as expected from the Ritter method.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of CRT-D SonR system as compared to SoC programming methods to:

* Increase the rate of patients responding to CRT
* Provide appropriate hemodynamic cardiac effect, as expected from the Ritter method.

The identification of CRT responders, as defined by echocardiography, generally refers to a significant reduction of the LV End-Systolic Diameter (LVESD) and/or LVESV during Follow-Up (FUp).

Patients will be considered as responders to CRT if their LVESV decreased by > 15% after 6 months of CRT therapy as compared to baseline. The percentage of CRT responders will be compared between the two study arms.

SoC is defined as the standard CRT system programming/optimization method currently used by physicians in study centers and any method may be used in the study if considered as routine practice in the study center.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for implantation of a CRT-D device according to published relevant ESC and CCS guidelines ;
* In Sinus Rhythm;
* Have reviewed, signed and dated an informed consent

Exclusion Criteria:

* Previous implant with a pacemaker, an Implantable Cardioverter-Defibrillator or a CRT device (except upgrade from single chamber ICD with a fully functional defibrillation lead not under recall or surveillance);
* Persistent atrial arrhythmias (or cardioversion for Atrial Fibrillation) within the past month;
* Ventricular tachyarrhythmia secondary to reversible causes such as acute myocardial infarction (MI), digitalis intoxication, drowning, electrocution, electrolyte imbalance, hypoxia or sepsis, uncorrected at the time of the enrolment;
* Incessant ventricular tachyarrhythmia;
* Unstable angina, or acute MI, Coronary Artery Bypass-Grafting (CABG), or Percutaneous Transluminal Coronary Angioplasty (PTCA) within the past 4 weeks;
* Correctable valvular disease that is the primary cause of heart failure;
* Mechanical heart valve or indication for valve repair or replacement;
* Recent Cerebro-Vascular Accident (CVA) or Transient Ischemic Attack (TIA) (within the previous 3 months);
* Post heart transplant (patients who are waiting for a heart transplant are allowed in the study);
* Already included in another clinical study that could confound the results of this study;
* Life expectancy less than 1 year;
* Inability to understand the purpose of the study;
* Unavailability for scheduled follow-up or refusal to cooperate;
* Sensitivity to 1 mg Dexamethasone Sodium Phosphate (DSP);
* Age of less than 18 years;
* Pregnancy;
* Drug addiction or abuse;
* Under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
CRT-responders rate increase based on LVESV decrease at M6 / baseline | 6 months
  For the purpose of this study, CRT-responders are defined as patients experiencing a decrease in LVESV of 15% or more at M6 Fup as most clinical trials used.
  The main objective of the SONR-ECHO trial is to show a minimum increase of CRT-responders rate of 15% (up to 72% or more) in the SonR study group as compared to SoC arm.

SECONDARY OUTCOMES:
A-wave truncation assessment at M6 | 6 months
  The Ritter's method attempts to optimize AV and VV timings in dual-chamber PM patients. According to this method, AV delay is optimal when LVFT is maximal and mitral valve closure only occurs after atrial systole (A-wave) is complete.

OTHER OUTCOMES:
Report LV remodeling from LVEDV decrease at M6 / baseline | 6 months
  LVEDV is a standard marker of CRT effectiveness. Echocardiographic data collected at M6 FUp will document the evolution of LVEDV as compared to baseline in order to assess CRT effectiveness.
LVEF increase at M6 | 6 months
  LVEF, as a surrogate of LVESV and LVEDV, is a standard marker of CRT effectiveness. Echocardiographic data collected at M6 FUp will document the evolution of LVEF as compared to baseline in order to assess CRT effectiveness.
AF analysis during FUp | 6 months
  Sorin commercialized CRT-D device offering both SonR optimization algorithm and atrio biventricular provides a performing Mode Switch (MS) function able to store and document sustained AF episodes during FUp.
  The MS data stored inSorin commercialized CRT-D device offering both SonR optimization algorithm and atrio biventricular memories will be collected at each FUp in order to report total AF burden, permanent AF and AF event free-rate in both arms up to M6 FUp.
AF-related events | 6 months
  Number of AF-events per patients, the event type, time to the first occurrence, the survival (event-free) curves will be reported per study group.
LA and RV functions | 6 months
  Echocardiographic data from each exam will be analyzed in order to report the evolution of the diastolic and systolic functions of the LA and of the RV per study group.
Adverse events | 6 months
  All AEs observed during FUp in all study patients will be classified by origin, symptoms, severity, treatment and outcome per study arm.

CONTACTS AND LOCATIONS:
Overall Officials: François Philippon, Principal Investigator — Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ)
Locations (1):
- Institut universitaire de Cardiologie et Pneumologie de Québec, Québec, Canada